CLINICAL TRIAL: NCT03225404
Title: Effectiveness of Percutaneous Electrolysis in the Treatment of Lateral Epicondylalgia. A Single-Blind Randomized Controlled Trial.
Acronym: MRH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cadiz (Other)
Responsible Party: Principal Investigator, Manuel Rodriguez Huguet, Clinical Professor, University of Cadiz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCadiz
Record Dates: First submitted 2017-07-17; First posted 2017-07-21 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Epicondylitis
Keywords: Tendinopathy; Electrolysis; Exercise; Dry needing
MeSH Terms: conditions — Tendinopathy; Motor Activity

STUDY DESIGN:
Intervention Model Description: A specialist physician will be diagnosed the epicondylitis
Who Masked: Participant
Masking Description: Outcomes assesor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): EPTE + EXER Therapeutic Percutaneous Electrolysis once week for four weeks associated with eccentric exercises devices at home.
  Interventions: Other: Epte group
- Control group (Experimental)
  Interventions: Other: Dry needling group

INTERVENTIONS:
Other: Epte group — Therapeutic Percutaneous Electrolysis once week for four weeks associated with eccentric exercises devices at home.
  Other Names: EPTE + EXER
  Arms: Experimental group
Other: Dry needling group — The intervention for this group consisted of dry needling in trigger points associated with eccentric exercises devices at home.
  Other Names: DN +EXER
  Arms: Control group

SUMMARY:
The concept of epicondylitis refers to the manifestation of pain ni the area of insertation of the epicondile muscles, and that it is accompained by limitation funcional.A tendinopathy is characterized as a process of degenaration, with fibroblast proliferation and disorganization of the fibers of collagen. This tendon pathology especially affects the epicondyle extensors and especially the first and second radial and short extensor carpal.

DETAILED DESCRIPTION:
Eccentric exercises of the epicondyle muscles were performed in 3 sets of 10 repetitions. Participants were asked to perform the exercise program on an individual basis twice every day for 4 weeks. The eccentric program consisted of 3 exercises, focusing on the epicondyle muscles. Participants were asked to do a normal flexion extension (concentric phase) and a slow return to the initial position (eccentric phase) included first the concentric phase, and the eccentric phase was slowly conducted. The exercise program was taught by a physiotherapist in the first session and monitored in the subsequent sessions.

ELIGIBILITY:
Inclusion criteria:

- Patients of both sexes, aged between 18 and 60 years, in an active state of pain and with a diagnosis of one month of evolution.

Exclusion Criteria:

- Patients who are pregnant, have pacemakers and those surgically operated patients who have been treated with Epte a month earlier

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2018-08-18 (Actual); Study Completion 2018-09-18 (Actual)

PRIMARY OUTCOMES:
The intensity of pain in epicondylitis | Baseline
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) will be used to assess the patients' current level of elbow pain, and the worst and lowest level of pain experienced in the preceding week in the elbow area.

SECONDARY OUTCOMES:
The intensity of pain in epicondylitis | Four and twelve weeks
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) will be used to assess the patients' current level of elbow pain, and the worst and lowest level of pain experienced in the preceding week in the elbow area.
Active elbow range of motion | Baseline,four and twelve weeks
  Measured by a two branches egoniomter
Pressure pain thresholds in epicondylitis trigger points | Baseline, four and twelve weeks
  Pressure pain thresholds (PPTs) will be measured with a pressure algometer (Baseline)
Questionnaire SF 12 | Baseline,four and twelve weeks
  The multidimensional health related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Rodriguez Huguet, Physiotherapy, Principal Investigator — University of Cadiz
Locations (1):
- Policlínica Santa maría, Cadiz, Cádiz, Spain

REFERENCES:
- [Background] Valera-Garrido F, Minaya-Munoz F, Medina-Mirapeix F. Ultrasound-guided percutaneous needle electrolysis in chronic lateral epicondylitis: short-term and long-term results. Acupunct Med. 2014 Dec;32(6):446-54. doi: 10.1136/acupmed-2014-010619. Epub 2014 Aug 13. PMID 25122629
- [Background] Minaya-Munoz F, Medina-Mirapeix F, Valera-Garrido F. Quality measures for the care of patients with lateral epicondylalgia. BMC Musculoskelet Disord. 2013 Oct 30;14:310. doi: 10.1186/1471-2474-14-310. PMID 24172311
- [Background] Mintken PE, Glynn P, Cleland JA. Psychometric properties of the shortened disabilities of the Arm, Shoulder, and Hand Questionnaire (QuickDASH) and Numeric Pain Rating Scale in patients with shoulder pain. J Shoulder Elbow Surg. 2009 Nov-Dec;18(6):920-6. doi: 10.1016/j.jse.2008.12.015. Epub 2009 Mar 17. PMID 19297202
- [Background] Arias-Buria JL, Truyols-Dominguez S, Valero-Alcaide R, Salom-Moreno J, Atin-Arratibel MA, Fernandez-de-Las-Penas C. Ultrasound-Guided Percutaneous Electrolysis and Eccentric Exercises for Subacromial Pain Syndrome: A Randomized Clinical Trial. Evid Based Complement Alternat Med. 2015;2015:315219. doi: 10.1155/2015/315219. Epub 2015 Nov 15. PMID 26649058